CLINICAL TRIAL: NCT03153787
Title: Influence of Vaginal and Endometrial Microbiome on the Results of Assisted Reproduction Techniques and Probiotic Administration Effect: Controlled Before-and-after Study
Brief Title: Vaginal Microbiome Influence on the Results of Assisted Reproduction Techniques
Acronym: RIFMicrobiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Andrea Bernabeu García, Principal Investigator, Instituto Bernabeu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Microbioma2017
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Implantation Failure
Keywords: implantation failure; fertility; microbiome; Assisted reproduction
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Not pregnancy (Experimental): Vaginal probiotic administration
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic — Vaginal probiotic administration according to the standard regimen: 1 tablet (via vaginal) for 5 days after menstruation during the same cycle of the next embryo transfer.

SUMMARY:
The objective of the present study to analyze the vaginal microbiome in patients who have not achieved gestation after oocyte donation treatment and after probiotic administration.

All patients will receive vaginal probiotic according to the standard regimen. Sample collection will be performed the embryo transfer day and on the day of the pregnancy test. Follow up of gestation will be carried out.

The analysis of the vaginal microbiome will be performed though massive genetic sequencing (determination of 16SRNA).

The study variables, among others, are vaginal microbiome pattern after probiotic administration, the gestation rate, and the abortion rate.

DETAILED DESCRIPTION:
This study will be performed after the observational study "Vaginal microbiome influence on the results of assisted reproduction techniques". The main goal of this previous study will be to identify patterns of vaginal and / or endometrial microbiome in relation to the gestation rate in women with implantation failure and / or repeat abortions who undergo an oocyte donation treatment. The vaginal and endometrial microbiome of women with (i) implantation failure, (ii) repeat abortions and (iii) control group without implantation failure or repeat abortions, will be analyzed before and after the embryo transfer.

Those women who do not achieve pregnancy will be eligible for the present study. The objective of the present study to analyze the vaginal microbiome in patients who have not achieved gestation after oocyte donation treatment and after probiotic administration.

All patients will receive vaginal probiotic according to the standard regimen: 1 tablet (via vaginal) for 5 days after menstruation during the same cycle of the next embryo transfer.

The vaginal sample will be analyzed after taking the probiotic. Sample collection will be performed the embryo transfer day and on the day of the pregnancy test. Follow up of gestation will be carried out.

Vaginal sample collection: obtention of vaginal fluid with vaginal swab by direct visualization. Direct visualization means having the patient in a lithotomy position, like a routine gynecological examination by visualization with a vaginal speculum.

The analysis of the vaginal microbiome will be performed though massive genetic sequencing (determination of 16SRNA). First of all, the extraction of RNA and subsequent analysis. We will analyze the groups of microorganisms, as well as the determination of patterns related to failure of implantation, repetitive abortions and gestation success.

The study variables, among others, are vaginal microbiome pattern after probiotic administration, the gestation rate, and the abortion rate. The vaginal microbiome will be compared with the results of the previous observational study.

ELIGIBILITY:
Inclusion Criteria:

* Treated by oocyte donation.
* Transfer of a single euploid embryo in the blastocyst phase.
* <3 months prior without antibiotic treatment.
* Women who have completed the previous observational study "Study of the influence of vaginal and endometrial microbiome on the results of assisted reproduction techniques".
* Women who have not achieved gestation after treatment.
* Signed informed consent form.

Exclusion Criteria:

* Uterine malformations.
* Not treated hydrosalpinx
* Known factors of implantation failure and repetitive abortions, such as haematological disorders of hypercoagulability.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Vaginal microbiome at 2 and 4 weeks | 2 weeks and 4 weeks
  Vaginal microbiome will be analyzed through massive genetic sequencing (determination of 16S RRNA) Before and after probiotic administration
Gestation rate | 4 weeks
  Gestation rate after assisted reproduction technique
Abortion rate | 45 weeks
  Abortion rate (clinical and biochemical) after assisted reproduction technique

SECONDARY OUTCOMES:
Live newborn rate | 45 weeks
  Live newborn rate after assisted reproduction technique
Complications during gestation | 45 weeks
  Complications during gestation after assisted reproduction technique

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No